CLINICAL TRIAL: NCT06734364
Title: Functional Treatment of Non-thumb Metacarpal Shaft Fractures. Randomized Study Evaluating Buddy Taping Versus Splint on Functional Recovery of the Hand
Brief Title: Buddy Tape vs. Splint for Metacarpal Shaft Fracture Recovery
Acronym: SYNATIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A02344-43
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Non-thumb Metacarpal Shaft Fracture
Keywords: Metacarpal shaft fracture
MeSH Terms: interventions — Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- buddy (Experimental)
  Interventions: Device: buddy tape
- splint (Active Comparator)
  Interventions: Device: splint

INTERVENTIONS:
Device: buddy tape — Buddy-taping a finger dynamically splints one finger to an adjacent, uninjured finger.
  Arms: buddy
Device: splint — Short arm splint immobilize and maintain stability of the injured finger, the hand is immobilized in the intrinsic plus position with syndactyly of the injured finger and adjacent finger
  Arms: splint

SUMMARY:
The goal of this clinical trial is to see if buddy tape can treat shaft fracture of hand long fingers as well as splint.

The main question it aims to answer is: Two months after the fracture, are the hand activities as good with buddy taping as with splint? Researchers will compare buddy tape group to splint group to see if the strength of the arm is not lower with buddy tape.

Participants will attend 4 visits after receiving either buddy tape or splint, to control their hand strength and the correct healing of their franture.

DETAILED DESCRIPTION:
Patients will be identified in the emergency ward after x-rays are positive for a non-thumb metacarpal fracture. If they consent to participate in the study, they will be put into either the buddy taping or the short arm splint group. This decision will be made through randomization, and the physician will not select which group the patient is in.

As in routine practice, the patients are seen again on D15 ± 3 days, D30 ± 5 days and D60 ± 5 days in an orthopedic consultation with X-ray to control the hand face, strict profile and 3/4. Both devices are removed at the check-up consultation on day 30 ± 5 days.

The patients will then attend the end of trial visit at Day 90 ± 5 days in an orthopedic consultation with X-ray.

No specific act is added by this research.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient
2. Fingers 2 to 5 metacarpal shaft fracture, little or no displacement
3. Tilt less than or equal to thirty degrees
4. No rotation disorder
5. Patient who has given consent to participate in the study and has signed an informed consent

Exclusion Criteria:

1. Surgical treatment indicated
2. Patient pregnant or likely to be pregnant
3. Patient who does not speak or understand French
4. Subject under guardianship or curatorship
5. Subject not beneficiary of a social security system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2027-02-05 (Estimated)

PRIMARY OUTCOMES:
Quick Dash | day 60
  Auto questionnaire evaluating the disabilities of the arm, shoulder and hand

SECONDARY OUTCOMES:
clamp force | day 0,15,30,60 and 90
  Clamp force deficit measured by a hydraulic hand dynamometer
Grip force | day 0,15,30,60 and 90
  Grip force deficit measured by a hydraulic hand dynamometer
TPM | day 0,15,30,60 and 90
  Total passive motion measured with a digital goniometer
TAM | day 0,15,30,60 and 90
  Total active motion measured with a digital goniometer

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No